CLINICAL TRIAL: NCT06224400
Title: A Phase 1, First-in-Human, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Escalating Single and Multiple Doses of ENC1018 in Healthy Adult Subjects
Brief Title: A First-in-Human SAD/MAD Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ENC1018 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EnnovaBio Australia Pharmaceuticals Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: EnnovaBio (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENC1018-P1-01
Record Dates: First submitted 2024-01-08; First posted 2024-01-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ENC1018 for SAD (Experimental): 6 of out 8 subjects per cohort will be randomized to receive ENC1018
  Interventions: Drug: ENC1018 for SAD
- Placebo for SAD (Placebo Comparator): 2 of out 8 subjects per cohort will be randomized to receive placebo
  Interventions: Drug: Placebo for SAD
- ENC1018 for MAD (Experimental): 6 of out 8 subjects per cohort will be randomized to receive ENC1018
  Interventions: Drug: ENC1018 for MAD
- Placebo for MAD (Placebo Comparator): 2 of out 8 subjects per cohort will be randomized to receive placebo
  Interventions: Drug: Placebo for MAD

INTERVENTIONS:
Drug: ENC1018 for SAD — SAD: Healthy subjects meeting eligibility criteria will be sequentially randomized to each dose cohort (cohort A1-A6) to receive either ENC1018 or placebo. The investigational product (ENC1018 or placebo) will be administered orally as a single dose.
  Arms: ENC1018 for SAD
Drug: Placebo for SAD — SAD: Healthy subjects meeting eligibility criteria will be sequentially randomized to each dose cohort (cohort A1-A6) to receive either ENC1018 or placebo. The investigational product (ENC1018 or placebo) will be administered orally as a single dose.
  Arms: Placebo for SAD
Drug: ENC1018 for MAD — MAD: Healthy subjects meeting eligibility criteria will be sequentially randomized to each dose cohort (cohort B1-B3) to receive either ENC1018 or placebo. The investigational product (ENC1018 or placebo) will be administered orally for a total of 14 days.
  Arms: ENC1018 for MAD
Drug: Placebo for MAD — MAD: Healthy subjects meeting eligibility criteria will be sequentially randomized to each dose cohort (cohort B1-B3) to receive either ENC1018 or placebo. The investigational product (ENC1018 or placebo) will be administered orally for a total of 14 days.
  Arms: Placebo for MAD

SUMMARY:
This is a Phase 1, FIH, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, and PK characteristics of ENC1018 after single and multiple oral dose administration in healthy adult subjects.

The study will be conducted in two parts: Part A -Single ascending Dose (SAD) and Part B - Multiple ascending dose (MAD). A Food Effect Cohort will be conducted within Part A. Part A is for the single dose use of IP, while Part B is once daily use for 14 consecutive days.

Approximately 72 healthy adult subjects are planned to be enrolled. Each subject will be enrolled in only one cohort of either Parts A or B of the study, to receive only one dose regimen during the study. Part B may be initiated in parallel or prior to completion of Part A, at the discretion of Safety Review Committee (SRC), upon reviewing safety and plasma PK data.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects of any ethnic origin, must be between 18 and 55 years of age inclusive.
* Subject is in generally good health according to the Investigator's assessment as determined by medical history, physical examination, vital sign assessment, 12-lead ECG, and clinical laboratory evaluations.
* Subject has a negative urine drug screen, cotinine screen, and alcohol breath test.
* Nonsmoker
* Subject has Body Mass Index 18.0 to 32.0 kg/m2 inclusive, and body weight from 50 - 100 kg for male subjects, 45 -100 kg for female subjects
* Apply contraception methods for child-bearing potential subjects.

Exclusion Criteria:

* Have clinically relevant medical history or unstable hepatic, pulmonary, hematologicalor immunological disease making implementation of the protocol or interpretation of the study results difficult, or that would put the subject at risk by participating in the study, under the discretion of the Investigator.
* Any disease or surgical procedure (including cholecystectomy) that may substantially affect IP absorption, distribution, metabolism, and excretion as judged by the Investigator
* Any current active infections, including localized infections, or any recent history (within 1 week prior to IP administration) of active infections, cough, or fever; or a history of recurrent or chronic infections.
* Dosing with any other investigational drug or therapy within 90 days prior to dosing.
* Is positive for HBsAg,HCVAb, HIVAb, or tuberculosis.
* Pregnant, breast-feeding and/or lactating women
* Have received any live vaccines (bacterial or viral) within 12 weeks prior to Screening or intend to receive a live vaccine during the study period or within 30 days after the last dose of the IP.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Number and type of treatment emergent adverse events (TEAE) following ENC1018 administration will be assessed using the latest version of Medical Dictionary for Regulatory Activities (MedDRA 25.0 or above) | Day 1 through Day 8 (SAD) or 21 (MAD)
Severity of TEAEs following ENC1018 administration will be assessed using categories as mild, moderate and severe | Day 1 through Day 8 (SAD) or 21 (MAD)
Evaluations of clinical laboratory and changes from baseline will be assessed using descriptive statistics following ENC1018 administration | Day 1 through Day 8 (SAD) or 21 (MAD)
  Laboratory values include hematology, biochemistry, clinical chemistry, coagulation, and urinalysis
Evaluations of physical examinations and changes from baseline will be assessed using descriptive statistics following ENC1018 administration | Day 1 through Day 8 (SAD) or 21 (MAD)
  Physical examination include assessments of the skin, cardiovascular, respiratory, gastrointestinal, and neurological systems
Evaluations of vital signs and changes from baseline will be assessed using descriptive statistics following ENC1018 administration | Day 1 through Day 8 (SAD) or 21 (MAD)
  Vital signs include body temperature, respiratory rate, blood pressure, and pulse
Evaluations of 12-lead ECGs and changes from baseline will be assessed using descriptive statistics following ENC1018 administration | Day 1 through Day 8 (SAD) or 21 (MAD)
  ECG parameters include heart rate, PR interval, QRS duration, QT interval, and QTcF interval

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | SAD: Up to Day 4, 72 hours post dose; MAD: up to Day 17, 72 hours post last dose
Area under the plasma concentration versus time curve (AUC) | SAD: Up to Day 4, 72 hours post dose; MAD: up to Day 17, 72 hours post last dose
Time to maximum concentration (Tmax) | SAD: Up to Day 4, 72 hours post dose; MAD: up to Day 17, 72 hours post last dose
Terminal elimination half-life (t1/2) | SAD: Up to Day 4, 72 hours post dose; MAD: up to Day 17, 72 hours post last dose
Apparent oral plasma clearance (CL/F) | SAD: Up to Day 4, 72 hours post dose; MAD: up to Day 17, 72 hours post last dose
Apparent volume of distribution during the terminal phase (Vz/F) | SAD: Up to Day 4, 72 hours post dose; MAD: up to Day 17, 72 hours post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Philip Ryan, Doctor, Principal Investigator — Nucleus Network Pty Ltd.
Locations (1):
- Nucleus Network Pty Ltd., Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No